CLINICAL TRIAL: NCT05757271
Title: Serum Levels of Klotho as a Possible Biomarker of Peripheral Artery Disease Progression
Brief Title: Serum Levels of Klotho as a Possible Biomarker of Peripheral Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Flex Andrea, MD, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 2753
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Peripheral Arterial Disease
Keywords: Klotho; FGF23; MALE; MACE
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Klotho, a membrane-bound protein co-receptor for fibroblast growth factor 23 (FGF23), is involved in atherosclerotic process and cardiovascular diseases. It regulates blood glucose and cholesterol levels. In addition, the lack of klotho has been associated with endothelial dysfunction, calcification and accumulation of cholesterol in the arteries, leading to coronary heart disease.

The goal of this observational study is to evaluate the potential use of circulating klotho and FGF23 serum levels as biomarkers of major adverse limb events (MALE) and major adverse cardiovascular events (MACE) in patients with peripheral artery disease (PAD) and chronic limb threatening ischemia (CLTI) requiring a procedure of endovascular revascularization.

The main questions it aims to answer are:

* association between klotho and FGF23 serum levels and major adverse limb events (MALE) after lower extremity revascularization.
* association between klotho and FGF23 serum levels and major adverse cardiovascular events (MACE) after lower extremity revascularization.

Patients with PAD and CLTI requiring lower extremity endovascular revascularization will undergo blood sampling for the dosage of circulating klotho and FGF23 before the endovascular procedure.

Incidence of MACE and MALE will be collected in a 12-months follow-up and will be associated with klotho and FGF23 serum levels at baseline.

ELIGIBILITY:
Inclusion Criteria:

* age of at least 40 years
* Ankle/Brachial Index (ABI) of less than 80
* at least one lower limb stenosis greater than 50% documented by Ultrasound Color Doppler (US)
* stage 4 or 5 PAD diagnosis according to the Rutherford classification
* presence of chronic limb threatening ischemia
* indication for LER of the target arterial stenosis

Exclusion Criteria:

* pregnancy
* acute infections at present or in the previous month
* primary hyperparathyroidism
* revascularization of the lower limb in the previous 3 months
* diabetic foot ulcers with signs of active infection or osteomyelitis
* diabetic peripheral neuropathy
* homozygous familial hypercholesterolemia
* absolute contraindication to antiplatelet therapy
* thrombophilia
* active cancer
* active autoimmune disease
* liver disease at functional status B or C according to Child-Pugh
* contraindication to endovascular revascularization
* organ transplantation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll consecutive subjects with PAD and CLTI requiring for endovascular revascularization and admitted to Internal Medicine Cardiovascular Unit of the Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma.
Sampling Method: Probability Sample
Enrollment: 207 (Estimated)
Dates: Start 2019-10-23 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Association between incidence of MALE and klotho and FGF23 serum levels | 12-months follow-up
  To evaluate the association between klotho and FGF23 serum levels before endovascular revascularization and MALE during the follow-up period.

SECONDARY OUTCOMES:
Association between incidence of myocardial infarction and klotho and FGF23 serum levels | 12-months follow-up
  To evaluate the association between klotho and FGF23 serum levels before endovascular revascularization and myocardial infarction during the follow-up period.
Association between incidence of stroke and klotho and FGF23 serum levels | 12-months follow-up
  To evaluate the association between klotho and FGF23 serum levels before endovascular revascularization and stroke during the follow-up period.
Association between incidence of cardiovascular death and klotho and FGF23 serum levels | 12-months follow-up
  To evaluate the association between klotho and FGF23 serum levels before endovascular revascularization and cardiovascular death during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Flex Andrea, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy